CLINICAL TRIAL: NCT03243058
Title: A Randomized, Double Blind, Phase I/II Trial of Low-Dose Interlekin-2 Immunotherapy in Established Type 1 Diabetes
Brief Title: Low-dose IL-2 in Established T1D - The "PROREG" Study
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding withdrawal and COVID-19 environment.
Sponsor: Jay S. Skyler (Other)
Collaborators: Diabetes Research Institute Foundation (Other); University of Florida (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor-Investigator, Jay S. Skyler, Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20170301; 20170301 (Other: University of Miami Central IRB)
Record Dates: First submitted 2017-07-20; First posted 2017-08-08 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes; Diabetes, Autoimmune
Keywords: Diabetes; Type 1 Diabetes; Autoimmune; Diabetes, Autoimmune; Interleukin-2; Interleukin; IL-2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — aldesleukin; Interleukin-2

STUDY DESIGN:
Intervention Model Description: ILT-101 (aldesleukin; Interleukin-2, IL-2), 0.5 million IU (body surface area <2 m2) or 1 million IU (body surface area >2 m2), or placebo, will be given for 5 consecutive days (days 1-5), and then on day 15 and every 15 days thereafter, for one year; at the one-year endpoint, approximately half the subjects on ILT-101 will continue therapy and the other half will switch to placebo for 1 more year.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The randomization will be performed by the Coordinating Center at the University of Miami. The participants will not be informed regarding the intervention assignment until the end of the study. The investigators and clinic personnel will also be masked as to study assignment. Laboratories performing assays for this protocol will be masked as to the identity and group assignment of biological materials to be studied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Arm (Active Comparator): ILT-101 (Aldesleukin; IL-2), 0.5 million IU/m2 (up to a maximum of 1 million IU), or placebo, will be given for 5 consecutive days (days 1-5), and then on day 15 and every 15 days thereafter, for two years.
  Interventions: Biological: ILT-101 (Aldesleukin; IL-2)
- Treatment-Placebo Arm (Experimental): Participants in this group will receive study drug ILT-101 for one year, and then placebo for the second year.
  Interventions: Biological: ILT-101 (Aldesleukin; IL-2); Other: Treatment-Placebo Arm
- Placebo (Placebo Comparator): Participants in this group will receive a placebo injection for two years.
  Interventions: Other: Placebo Arm

INTERVENTIONS:
Biological: ILT-101 (Aldesleukin; IL-2) — Administration of Low-Dose Interleukin-2 (ILT-101) for two years
  Other Names: IL-2; Interleukin-2
  Arms: Treatment Arm; Treatment-Placebo Arm
Other: Treatment-Placebo Arm — Administration of Low-Dose Interleukin-2 (ILT-101) for one year, and then placebo for the second year.
  Arms: Treatment-Placebo Arm
Other: Placebo Arm — Participants in this group will receive a placebo injection for two years.
  Arms: Placebo

SUMMARY:
Randomized, controlled, double-blinded, multicenter, phase I/II clinical trial to evaluate the safety of low-dose IL-2 and determine whether low-dose IL-2 therapy for one year, can prevent further loss of beta-cell function in patients with established T1D, (primary outcome). The study will carefully examine various effects of low-dose IL-2 on the immune system in patients with T1D, including effects on Treg and other cell subsets, and disease-specific autoimmune responses.

DETAILED DESCRIPTION:
Randomized, controlled, double-blinded, multicenter, phase I/II clinical trial to evaluate the safety of low-dose IL-2 and determine whether low-dose IL-2 therapy for one year, can prevent further loss of beta-cell function in patients with established T1D, (primary outcome). The study will carefully examine various effects of low-dose IL-2 on the immune system in patients with T1D, including effects on Treg and other cell subsets, and disease-specific autoimmune responses.

Patients will be treated with ILT-101 or placebo. ILT-101 will be given at doses of 0.5 million IU (body surface area <2 m2) or 1 million IU (body surface area >2 m2), via subcutaneous (s.c.) injections. Patients will receive a course of 5 daily injections (days 1-5. Starting on day 15, patients will receive an s.c. injection (same dose) every 15 days for 1 year. Thus, patients will receive 29 injections during the first year of treatment. At the end of the first year, approximately half of those randomized to ILT-101 will continue receiving treatment every 15 days, until the end of the second year (23 doses). The other half will stop therapy and will be switched to a placebo.

A group of patients will be randomly assigned to a placebo for the duration of the study. Patients to be included in this study are those diagnosed with T1D who would have had T1D from 4 months to 1 year at the time of randomization, who have a current or past demonstration of autoimmunity (using autoantibodies), and maintain preserved β-cell function, defined as an MMTT stimulated C-peptide >0.2 nmol/L. This population is chosen because it will extend the scope of therapy beyond the immediate time following diagnosis when most previous studies of immunotherapy in T1D have been conducted. This trial can further impact the field if a therapeutic benefit is shown when the disease is more established.

ELIGIBILITY:
Inclusion Criteria:

* 8-21 years of age
* T1D, demonstrated by at least one islet autoantibody
* T1D duration 4-12 months at the time of the first dose
* Peak stimulated C-peptide >0.2 nmol/L during a 4-hour MMTT

Exclusion Criteria:

* Treatment with oral anti-diabetic agents
* Illnesses that would preclude use of low-dose IL-2

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
C-peptide response | 1 year primary outcome
  Preservation of insulin secretion (measured as c-peptide nmol/L) based on stimulated area under the curve (AUC) during a 4-hour MMTT at 1 year

SECONDARY OUTCOMES:
C-peptide response | 2 year secondary outcome
  Preservation of insulin secretion (measured as c-peptide nmol/L) based on stimulated area under the curve (AUC) during a 4-hour MMTT at 2 years

OTHER OUTCOMES:
Proportions of regulatory T cells at (a) 1 year, (b) 2 years | 1 Year and 2 Years
Changes in insulin requirements | 1 Year and 2 Years
HbA1c level | 1 Year and 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Jay S Skyler, M.D., Principal Investigator — Professor of Medicine; Alberto Pugliese, M.D., Principal Investigator — Professor of Medicine; David A Baidal, M.D., Principal Investigator — Assistant Professor of Medicine
Locations (1):
- Diabetes Research Institute, University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
A participant's privacy and confidentiality will be respected throughout the study. Each participant will be assigned a unique identification number and these numbers rather than names will be used to collect, store, and report participant information. Site personnel will not transmit documents containing personal health identifiers (PHI) to the study sponsor or their representatives.